CLINICAL TRIAL: NCT05323513
Title: The Correlation Between Luteal Serum Progesterone and Live Birth Rate in IVF - a Prospective Cohort Study (LUT-2)
Brief Title: The Correlation Between Luteal Serum Progesterone and Live Birth Rate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peter Humaidan (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Other Study IDs: LUT-2
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study design is an observational cohort study. Level of serum P4 will be collected on day OR+4 as well as on the day of embryo transfer (ET) either day OR+3 or OR+5.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* BMI <35kg/m2

Exclusion Criteria:

* No fresh embryo transfer
* Prior participation in the study

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients treated at The Fertility Clinic, Regional Hospital in Skive, who meets the inclusion criteria will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate in relation to luteal serum progesterone levels on day four and three or five | 9-24 months after inclusion
  The birth of a live born child after gestational week 22+0

SECONDARY OUTCOMES:
Pregnancy rate in relation to luteal serum progesterone levels | 14-16 days after oocyte retrieval
  Serum Human chorionic gonadotropin<10 IU/l
Clinical pregnancy rate in relation to luteal serum progesterone levels | 7-9 weeks after inclusion
  Ultrasound scan detection of intrauterine fetal heartbeat in gestational week 7-9

CONTACTS AND LOCATIONS:
Overall Officials: Peter Humaidan, Professor, Principal Investigator — Fertilitetsklinikken, Regionshospitalet Skive
Locations (1):
- Fertilitetsklinikken, Regionshospitalet Skive, Skive, Denmark

IPD SHARING:
Plan to Share IPD: Undecided